CLINICAL TRIAL: NCT00881244
Title: Phase I Open Label Study of AS1411 in Advanced Solid Tumours
Brief Title: Study of AS1411 in Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Chris Smyth, VP Clinical Operations, Antisoma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS1411-C-101
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — AGRO 100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AS1411
  Interventions: Drug: AS1411

INTERVENTIONS:
Drug: AS1411 — I.v. 4-7 days, 1-40 mg/kg/day

SUMMARY:
A Phase I open label study of AS1411 in advanced solid tumours. Objectives include determining the MTD and DLT of AS1411, to determine the PK profile of AS1411 and to obtain preliminary evidence of clinical and biological responses to AS1411 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumours that were refractory to conventional/standard treatment
* Age >/ 18 years
* ECOG performance status </ 2 (Karnofsky >/60%
* Life expectancy >/ 8 weeks
* Adequate organ and marrow function

Exclusion Criteria:

* Radiotherapy or chemotherapy in the 4 weeks before study entry (6 weeks for nitrosourea or mitomycin C
* Lack of recovery from adverse events (AEs) caused by agents administered before study entry; current use of other investigational agent(s)
* Uncontrolled brain metastases including a need for corticosteroid therapy
* Pregnancy
* Uncontrolled intercurrent illness
* Psychiatric illness/social situations that could limit compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of AS1411

SECONDARY OUTCOMES:
To determine the pharmacokinetic (PK) distribution and profile of AS1411
To obtain preliminary evidence of clinical and biological responses to AS1411

CONTACTS AND LOCATIONS:
Locations (1):
- James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky, United States